CLINICAL TRIAL: NCT04035954
Title: Effects of Modified Pilates Exercises on Body Control, Gait and Function in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Hatice Adıgüzel, Principal Investigator, Sanko University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sanko University
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; modified pilates; trunk; gait; function; core stability
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study will include16 children with cerebral palsy (SP) diagnosed at the GMFCS I-II-III level with 8 controls and 8 treatment groups by random minimization between 7-14 years of age with 1 and 1+ spasticity on the lower extremity according to the Modified Ashworth Score.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Active Comparator): The control group will continue the routine physiotherapy program based on NDT: Neurodevelopmental Therapy twice a week, 2 days / 1 hour / day during 8 weeks.
  Interventions: Other: exercise
- Experimental (Experimental): The treatment group will participate in clinical pilates exercises 2 days / 1 hour / day during 8 weeks.They will also continue their weekly routine physiotherapy programs.
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — The control group will continue the routine NDT: Neurodevelopmental Therapy-based physiotherapy program twice a week. The treatment group will participate in clinical pilates exercises for 2 hours / day for 1 hour / 8 weeks. They will also continue their weekly routine physiotherapy programs.

SUMMARY:
Children with cerebral palsy (CP) have limitations in postural reactions and antigravity movements. Trunk control is the determinant of posture, balance, walking and functional activities. Core stability connects deep abdominal muscles, spine, pelvis, and shoulder girdle to protect the posture and provides support for extremity movements. Pilates and core stabilization were associated with postural control in elderly, MS and stroke individuals and it was concluded that pilates caused an increase in trunk stabilization. There are not enough studies investigating the effectiveness of pilates exercises in CP. The aim of this study was to investigate the effects of modified pilates exercises on body control, gait and functionality in children with CP.

DETAILED DESCRIPTION:
Postural control is the ability of the body to control its position in space for stability and orientation. Postural stability and balance are achieved by keeping the center of gravity of the body within the support surface. Stability can also occur with a static response when the body is stationary, and a dynamic response to internal or external perturbations when it is mobile. Antisipation of perturbation forces requires an effective core stabilization muscle activation as well as an effective integration of stimuli from different sensory systems. Trunk control is also provided by this relationship between neural systems and skeletal muscles. Children with CP show deficits in proximal muscle co-contraction and vertical posture stabilization, with limitations in postural reactions and antigravity movements. Trunk control is the determinant of balance, gait and functional activities from the early period. Core stability; it connects with deep abdominal muscles, spine, pelvis and shoulder girdle muscles to protect the posture and provide support for limb movement. During reaching out, stepping and sudden perturbations, the Transversus Abdominus muscle is activated primarily from other trunk and limb muscles, creating a core stability. Core activity includes not only spinal stability and power generation, but also many upper and lower extremity movements. Control is established by focusing on the transversus abdominis muscle by core stabilization training with Pilates, stabilization of trunk muscles. The proximal extremity muscles of the hip are also important to maintain the upright posture and maintain mobility. For example; hip abductor muscle strength compared to the knee and ankle muscles, walking variables and motor functions in children with CP were more correlated. Although the importance of walking was determined, activation patterns of trunk and hip muscles during walking were examined in a limited number of studies in individuals with CP. The effects of pilates on healthy adults, elderly, multiple sclerosis, stroke and musculoskeletal disorders were investigated and resulted in increased trunk stabilization.Therefore, it is thought that pilates can be applied in terms of muscle strength and postural control in children who can walk, stand independently, but need to develop some components for controlled movement. There are not enough studies investigating the effectiveness of pilates exercises in CP. The aim of this study was to investigate the effects of modified pilates exercises on body control, gait and function in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with CP at the level of GMFCS I-II-III between the ages of 5-18
* Not having any Btx / surgery in the last 6 months
* Lower extremity spasticity 1 and 1+ according to modified Ashworth score
* Signing the written informed consent form
* Who can follow verbal commands

Exclusion Criteria:

* Individuals with multiple disabilities (hearing, speaking, seeing)
* Individuals with any behavior disorder (Autism, etc.) / Mental problems
* Patients with congenital cardiorespiratory status
* Have received any specific core stabilization training over the last 6 months
* Mixed musculoskeletal / axial deformities

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Change of Prone Plank Test | first day of intervention and after the 8 weeks
  Its a core stability performance test. Patients are asked to raise their trunk by giving weight to the forearms and toes while the prone and elbows are in the flexion position.It meausures core stability in this position.Subjects will be encouraged to maintain the isometric postures for prone plank position as long as possible. The length of time subjects could maintain the correct position was recorded.The longest time of 2 trials, to the nearest 0.1 second, will be used for data analysis.
Change of Side Plank Test | first day of intervention and after the 8 weeks
  Its a core stability performance test. Patients are asked to raise their trunk by giving weight to the forearms and toes while the prone and elbows are in the flexion position.It meausures core stability in this position.Subjects will be encouraged to maintain the isometric postures side plank test position as long as possible. The length of time subjects could maintain the correct position was recorded.The longest time of 2 trials, to the nearest 0.1 second, will be used for data analysis.
Change of Modifiye Beiring Sorensen Test | first day of intervention and after the 8 weeks
  Tests the endurance capacity of posterior spinal musculature. The subject is positioning in prone lying position with pelvis at edge of the treatment table with the pelvis and legs well stabilized either manually. Initially the subjects supports their upper extremity on stool/bench in front of table until they are instructed to cross their arm and assume a horizontal position which is to be maintained as long as possible. Total time (in seconds) for which he/she was able to maintain horizontal position (i.e. the time between the assumption of the horizontal position up to the moment when they lost the horizontal position), was manually recorded using digital stopwatch up to two decimal places.
Change of Abdominal Fatigue test | first day of intervention and after the 8 weeks
  It measures the endurance of the anterior abdominal wall by asking the person to hold a sit- up position as long as they can. The subjects are required to sit on the test bench t and place the upper trunk against a support with an angle of 60 degree from the test bench. Both knee and hip are flexed to 90 degree .Both arms are folded across the chest with the hands placed on the opposite shoulder and toes are stabilized to the bed (either by manual support or by straps). The subjects are asked to maintain the body position while the supporting back support is withdrawn. The stopwatch is started at the moment, when the support is withdrawn. The stopwatch is stopping when the upper body fell below the 60 degree position.Time duration between these two points are recorded as the endurance holding score of the anterior abdominal muscle group.

SECONDARY OUTCOMES:
Change of Sharman's core stabilite testi (PBU=Pressure Biofeedback Unit Test) | first day of intervention and after the 8 weeks
  It is objective and clinically feasible method to evaluate core stability in the laboratory settings which uses a stabilizer Pressure Biofeedback Unit with its inflatable pad placed in the inflatable cell was placed centrally beneath the abdomen with the lower edge at the level of the anterior superior iliac spines while the subject is lying supine, and is inflated to certain pressure of 70 mm Hg.The person is asked to pull his belly in as much as he can in a tight pants. While this is observed, the development of any other movement strategy (breast swelling, breath holding, pelvis movement) is noted and inhibited. The pressure may drop 6-10mmHg from the limit line. After the start, the test is terminated when 10 repetitions and 10 seconds of contraction are formed. Times are measured with a stopwatch. At each contraction, the onset of PBU is 70 mmHg, pressure changes and averages after 10 contraction are calculated. No feedback is given to the patient during the measurement.
Change of Sit Ups Test | first day of intervention and after the 8 weeks
  Its a core test of power. The patient is asked to perform trunk flexion while the knees are in the flexed position and the feet are stabilized.The number of sit ups it can perform in 30 seconds is recorded.
Change of Modified Push-ups Test | first day of intervention and after the 8 weeks
  Its a core test of power. When the cases are in the prone position, the arms and elbows are asked to lift the head, shoulders, and trunk from the flexion with the elbows fully extended. During the test, the knees are positioned in flexion.The number of push ups it can perform in 30 seconds is recorded.
Change of 6 Minute Walk Test | first day of intervention and after the 8 weeks
  The 6-minute walk test (6MWT) is a standardized, self-paced walking test commonly used to assess functional ability in children with cerebral palsy (CP).1 The test has been reported to reflect functional capacity in terms of activities of daily living.2 In a recent Delphi study3 surveying the views of 15 physical therapy and exercise physiology experts, the 6MWT has been recommended as a submaximal exercise test for children with CP of Gross Motor Function Classification System4 (GMFCS) levels I to III.
Change of Pediatric Reach Test (PRT) | first day of intervention and after the 8 weeks
  PRT was developed and modified from Functional Reach Test which was originally developed for measuring standing functional reach in adult populations. Due to the consideration that many children with CP are only able to maintain the upright position in sitting, PRT is developed to measure the maximal reach distance of children with CP both in sitting and standing positions. The total score of PRT is the sum of scores of PRT during sitting and PRT during standing.
Change of Physician Rating Scale (PRS) | first day of intervention and after the 8 weeks
  One of these instruments is the Physician Rating Scale (PRS), an observational clinical evaluation of gait. This simple scale records gait in the sagittal plane only. Gait variables are recorded in the subtitle of Crouch, Knee, Foot contact scoring and general Change. Several items are geared to quantify visually the relationship between the ankle and knee position during stance. Maximum total score is 10.Also maximum scores shows the better results.
Change of Berg Balance Scale (BBS) | first day of intervention and after the 8 weeks
  The BBS is a simple measure with 14 items that can be completed within 20 minutes. These items are used to test functional skills relevant to everyday tasks, progressing from stable positions to position changes and finally to the upright position with various maneuvers to challenge balance. The items are scored on a 5-point ordinal scale from 0 to 4 (0-1-2-3-4). The highest score is 56 points; a higher score indicates a better functional balance performance.
Change of Seated Postural Control Measure (SPCM) | first day of intervention and after the 8 weeks
  SPCM has two sections. One section examines postural alignment and consists of 22 items; the other section examines functional movement and consists of 12 items. The SPCM can be administered and scored in 20 minutes or less. An ordinal scale of 0 to 3 is used to score each segmental posture. A given deviation, whether to the right or the left, would receive the same score. Visual observation and palpation are the only methods used to estimate postural alignment. At the beginning of the assessment, the child is placed in the seat in what the assessing therapist considers an optimal position. Verbal encouragement (without manual support) to maintain a correct posture is given. Each of the items in the function section consists of four levels, with higher grades representing better task achievement (from zero to completion). A maximum of 1 minute is allowed for motivating the child and completing each item. If more than one attempt is made, the best performance is scored.
Change of Gross Motor Function Classification System (GMFCS) | first day of intervention and after the 8 weeks
  The GMFCS is a common classification system and is an evidence-based classification tool of five levels ranging from level I, which includes children with minimal or no disability with respect to community mobility, to level V, which includes children who are totally dependent on external assistance for mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Adıgüzel, PhD cd., Principal Investigator — Sanko University; Bülent Elbasan, Ass. Prof., Principal Investigator — Gazi University
Locations (1):
- Sanko University, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adiguzel H, Elbasan B. Effects of modified pilates on trunk, postural control, gait and balance in children with cerebral palsy: a single-blinded randomized controlled study. Acta Neurol Belg. 2022 Aug;122(4):903-914. doi: 10.1007/s13760-021-01845-5. Epub 2022 Jan 18. PMID 35040072